CLINICAL TRIAL: NCT04886141
Title: Virtual Reality and Pediatric Dentistry: An Interventional Study Examining Distraction Comparing Virtual Reality Goggles to Nitrous Oxide During Dental Procedures
Brief Title: Virtual Reality and Anxiety in Pediatric Dentistry
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Geisinger Clinic (Other)
Responsible Party: Principal Investigator, Gayatri Malik, Pediatric Dentist, Geisinger Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-0138
Record Dates: First submitted 2021-05-06; First posted 2021-05-13 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Pediatric Dentistry

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care treatment with Scales (No Intervention): Patients will receive the standard of care restorative procedure with the addition of the FLACC pain scale, Wong Baker FACES Pain rating and Houpt scale to create a baseline data of pain to compare with the experimental group.
- Virtual Reality Headset (Experimental): Instead of receiving the Nitrous that would be used to help calm patients during the standard of care restorative procedure. Patients will be given a the Oculus Quest 2 Virtual realty headset and a video will be played. The FLACC pain scale, Wong Baker FACES Pain rating and Houpt scale data will be collected to compare the patients pain level between the two groups.
  Interventions: Behavioral: Virtual Reality Headset

INTERVENTIONS:
Behavioral: Virtual Reality Headset — To determine if virtual reality headsets can reduce a patients pain level instead of using the standard Nitrous. This may provide a alternate to patients who cannot receive nitrous if pain or anxiety can be reduced effectively.
  Arms: Virtual Reality Headset

SUMMARY:
Two groups of pediatric patients between the ages of 4 to 12 years old will be examined in this study. The treatment group will receive dental treatment while wearing Virtual reality Headset. Control group will receive the standard of care dental treatment with under nitrous sedation. Procedures performed in all groups will be restorative treatments, which can include intraoral anesthetic injections, placing dental fillings, crowns, and the extractions of teeth. In group 1, A specific VR headset, the "Oculus Quest 2" will be used. Through the headset, a video will be played for the child during a dental procedure.

DETAILED DESCRIPTION:
This is a randomized controlled, interventional therapy utilizing virtual reality goggles as a method of distraction. Data will be collected during and after the procedure on the type of behavior displayed and the child's response to standardized questions. Pediatric patients aged 4-12 years who only require nitrous sedation to complete painful dental treatment which necessitates anesthesia will be included in this study. These patients exhibit Frankl 2-3 behavior, requiring behavior guidance in order to complete the procedure. Frankl 1 or 4 children, those who do not need behavior guidance at all, or children with heavy behavior guidance who would not be able to complete the procedure, will be excluded.

Participants will be recruited in the clinic, during a new patient exam, routine hygiene or operative dentistry appointment. Following the Frankl behavior score diagnosis, an evaluation of behavior will happen during the beginning of the appointment, specifically watching for acceptance of treatment plan, openness to conversation, and any defiant behaviors or crying. If the child had previously presented as Frankl 2-3 within 6 months of the day of screening, the child may be considered for the study.

The parent and child being recruited for the study will be informed of the nature of the study, the possible risks benefit and alternatives, and written consent will be obtained from the parent or legal guardian. Assent from child 7 to 12 will also be required as well. The qualifying patient will enter the operatory and be admitted into the study. Participants will be briefed on how the study will proceed, and will be randomized into a control group, (continuing a typical procedure using nitrous oxide ), or treatment group (continuing a procedure with the VR goggles). The groups will be selected at random prior to treatment in the study, using the flip of a coin. Both Groups will use of FLACC, Wong-Baker FACES, and Houpt Behavior scales to access the pain or discomfort of subjects. The treatment group will have the goggles placed on the head and in front of the eyes. The goggles are automatically set to start media as soon as the wearer dons them. The patient will be reclined, and placed in an ideal setting, and the goggles will be calibrated to the patient's current view. The dental procedure will then follow. Most procedures require a local anesthetic injection, and if the patient receives this injection, participants will be graded with FLACC score during the injection. At the end of the procedure the child will be evaluated using the Wong-Baker FACES scale, the Houpt Crying and Movement Scales, and a survey will be given to the patient to be completed.

Participants will participate in the study during a restorative dental appointment, however, some patients may need more the one restorative visit. Participants who require multiple restorative treatments will only being include in the study during one visit and no other research activities will occur after. Most appointments are projected to last a maximum of 1 hour. The limiting factor in all treatment in this study, will be the participant's willingness to participate in future appointments.

ELIGIBILITY:
Inclusion Criteria:

* Male or female pediatric dental patients age 4-12 years
* Require a restorative procedure that includes injection of anesthesia .
* Exhibiting behavior Frankel 2 or 3 during their new patient, recall or previous dental appointment.
* ASA 1 or 1

Exclusion Criteria:

* Children who exhibit behavior rated as Frankl 1, or Frankl 4.
* Have health issues that prevent use of VR Oculus headset,
* Hypersensitivity to audio-visual devices that can lead to seizures
* ASA 3 or 4

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 53 (Actual)
Dates: Start 2021-10-21 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-21 (Actual)

PRIMARY OUTCOMES:
Rate of effectiveness virtual reality goggles reduce pain | 12 months
  To determine if pain can be diminished or alleviated and if subjects had better cooperation or pain tolerance with the distraction through virtual reality headsets.

SECONDARY OUTCOMES:
Rate of effectiveness of virtual reality distraction to nitrous oxide | 12 months
  To determine if there is a difference in the effectiveness between the use of the standard nitrous oxide and VR distraction.

CONTACTS AND LOCATIONS:
Locations (1):
- Geisinger, Danville, Pennsylvania, United States